CLINICAL TRIAL: NCT02691520
Title: Epidemiology of Treatment Resistant Depression in Taiwan
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Elysia Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: CR108117; NOPRODDEP4001 (Other: Johnson & Johnson Pte Ltd)
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Taiwan Participants with Treatment Resistant Depression: Taiwan participants with Depression will be followed up to 8 years for incidence and duration of treatment resistant depression.

SUMMARY:
The purpose of this study is to assess the epidemiology of Treatment Resistant Depression (TRD) in the nationally insured population in Taiwan including incidence, duration of clinical episodes, and prevalence by age and sex.

DETAILED DESCRIPTION:
This is a retrospective study of approximately one million subjects randomly selected from an anonymized database National Health Insurance Research Database (NHIRD). Participants aged 18 years or older who have had neither a depression diagnosis nor a dispensing of an antidepressant medication in the last four months of 2004 will enter the study when they receive in 2005 a depression diagnosis and a dispensing of an antidepressant medication within 30 days of each other and will be followed up to 8 years or until they have 4 months with neither a depression diagnosis nor a dispensing of an antidepressant medication. Treatment Resistant Depression (TRD) Incidence, TRD prevalence by age and sex and duration of clinical episodes will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been continuously enrolled in the insurance plan since January 1, 2004 (ignoring breaks of less than 30 days) and have not received an exclusion diagnosis and during the last 4 months of 2004, a) Have not received a diagnosis of depression and b) Have not received a dispensing of an AD medication
* Participants with a diagnosis of a depressive disorder including dysthymic disorder (International Classification of Diseases [ICD]-9 codes 296 depression-related, 300.4, 311) and Major Depressive Disorder (ICD-9 296.2, 296.3) will be followed through December 31, 2013

Exclusion Criteria:

- Participants who receive following diagnosis will be excluded, a) Mania, b) Schizophrenia (ICD-9 codes 295), c) Bipolar disorder (ICD-9 codes 296 bipolar-related), D) Dementia (ICD-9 codes 290 or 294); Note: Major depressive disorder (MDD) with psychotic behavior (ICD 296.24 for single episode, ICD 296.34 for recurrent episode) is not an exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 and older are randomly sampled from the National Health Insurance Research Database (NHIRD).
Sampling Method: Probability Sample
Enrollment: 8356 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-18 (Actual)

PRIMARY OUTCOMES:
Incidence Percentage of Participants with Treatment Resistant Depression | Approximately 8 Years
  The percentage of beneficiaries of Taiwan's health insurance plan who developed treatment resistant depression during 2005
Prevalence Percentage of Participants with Treatment Resistant Depression | Approximately 8 Years
Duration of an episode of Depression | Approximately 8 Years
  Time from onset of depression to cessation of depression visits and medications.

SECONDARY OUTCOMES:
Healthcare costs | Approximately 8 Years
  Direct healthcare cost associated with depression treatment will be assessed.
Number of Participants With Comorbidities | Approximately 8 Years
Medications used by Participants with Treatment Resistant Depression | Approximately 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC